CLINICAL TRIAL: NCT05133960
Title: Validity and Reliability of the Activity Diversity Questionnaire for Turkish Older Adults
Brief Title: The Turkish Version of the Activity Diversity Questionnaire
Status: Completed | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Hasan Atacan Tonak, Asst. Prof. Dr., PT, PhD., Akdeniz University
Other Study IDs: ADQ
Record Dates: First submitted 2021-11-13; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Activity Diversity; Validity; Reliability; Older Adults; Outcome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire assessment — Validity and reliability of the Turkish Version of the Activity Diversity Questionnaire

SUMMARY:
The Activity Diversity Questionnaire (ADQ) was developed to assess activity diversity. The questionnaire consists of 20 items rated on a four-point Likert scale. This questionnaire defines activity diversity using Shannon's entropy and is the first assessment tool of activity diversity validated for validity and reliability. Important data can be obtained from this questionnaire, such as the relationship between the health status of older adults and their activity diversity. There is no scale in Turkish that can be used to evaluate the activity diversity. The aim of our study was to investigate the relevance of the Activity Diversity Questionnaire for Turkish older adults and the effectiveness of its clinical use.

DETAILED DESCRIPTION:
The Activity Diversity Questionnaire was developed by Junta Takahashi et al. in 2020 to assess activity diversity. The Activity Diversity Questionnaire was translated into Turkish using the back and forward translation method described by Beaton et al. First of all, the Activity Diversity Questionnaire, whose original text was in English, was translated into Turkish by 2 independent native speakers who have a good command of the culture of the scale and speak English very well. The scales translated from English to Turkish were analysed by another expert who knew English very well, and the translations were synthesized into a single translation. The Turkish synthesis translation of the Activity Diversity Questionnaire was translated back into English by 2 independent native speakers who are also familiar with Turkish culture and know Turkish very well. This phase was completed by people who were not related to the previous translation process and who had never seen the Activity Diversity Questionnaire before. The scales translated from Turkish to English were synthesized and turned into a single translation. This translation was emailed to Shuichi Obuchi, who developed the scale to avoid ambiguity. After obtaining confirmation from Shuichi Obuchi about the accuracy of the translation, the final version of the Turkish version of the Activity Diversity Questionnaire was reviewed, and the assessment of cultural adaptation and adaptation to the Turkish language was carried out by a Turkish linguist. After examining the compatibility of the translations, a pilot study was applied to 40 older adults in order to determine the clarity of the final version of the scale. The meaning of both the items and the responses was checked with the pilot assessment applied to the older adults. Participants completed the scale without any problems and the final version of the scale was created. Test-retest and internal consistency analyzes were applied to determine the reliability of the Activity Diversity Questionnaire. Confirmatory factor analysis with AMOS 26 was used to confirm the scale factors for construct validity analysis. After calculating the total scores obtained from all the scales applied for the criterion validity of the Activity Diversity Questionnaire, a comparison method with a previously validated scale was used using Spearman correlation analysis.

ELIGIBILITY:
Inclusion Criteria:

* ≥65 years
* MMSE (Mini-Mental State Exam) score ≥24
* being native language Turkish,
* having Turkish literacy skills,
* volunteering to participate in the study,
* having read and approved the informed consent form

Exclusion Criteria:

* Participants were asked, "Have you had any changes (eg, moving, feeling sick, traveling)?" in your life in the past week? Participants were asked to answer with "No change", "Small change" or "Major change". Participants who answered as "Major change" and had an MMSE <24 score were excluded from the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: 220 older adults aged ≥65 years, with Mini-Mental State Exam (MMSE) score ≥24, who did not experience any major changes in their life in the past week, were included in the study.
Sampling Method: Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Activity Diversity Questionnaire | 2 weeks
  The Activity Diversity Questionnaire was developed by Junta Takahashi et al. in 2020 to assess activity diversity. This scale is the first assessment tool of activity diversity validated for reliability and validity. The questionnaire consists of 20 items rated on a four-point Likert scale. Each item is scored using frequency scores ranging from 0 to 3 (0 = almost none, 3 = almost every day). In the Activity Diversity Questionnaire, the participants were asked the following question: "How many times have you done the following activities in the last week?" Each question was answered using a four-point Likert scale: "0: almost none", " 1: 1-2 days per week", "2: every 2 days" and "3: almost every day." Thus, frequency scores between 0 and 3 were assigned to each item. These frequency scores were then used to calculate a diversity score. As the score approaches 1, the activities diversity increases and diversity score are spread evenly across all 20 categories.
Barthel Activities of Daily Living Index | 1 week
  The Barthel index was developed by Mahoney and Barthel in 1965. The Turkish validity and reliability study of the Barthel Activities of Daily Living Index, which is simple, understandable and includes all the parameters of daily living activities, was conducted in 2000. The index consists of 10 subheadings: eating, bathing, self-care, dressing, bladder control, bowel control, toilet use, chair/bed transfer, mobility, and use of stairs. Its scoring ranges from 0-100. 0-20 points fully dependent, 21-61 points severely dependent, 62-90 points moderately dependent, 91-99 points mildly dependent, and 100 points complete independence.
Lawton Instrumental Activities of Daily Living Scale | 1 week
  The Lawton Instrumental Activities of Daily Living Scale was developed in 1969 by M. Powell Lawton and Elaine M. Brody. The Turkish validity and reliability study of the index, which was conducted in 2020, consists of a total of 8 questions that inquire about using the telephone, shopping, preparing food, cleaning the house, washing clothes, traveling by public transport or taxi, recognizing, and using medications and money management, which are necessary for living in society. Its scoring ranges from 0-8. Lower scores mean more dependence.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No